CLINICAL TRIAL: NCT05229445
Title: Safety of a Real-time Continuous Glucose Monitor-based Insulin Bolus Calculator: The "CGM-IBC" Study
Brief Title: A Continuous Glucose Monitor Based Insulin Bolus Calculator
Acronym: CGM-IBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Welldoc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WD001
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: continuous glucose monitor; insulin calculator
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single group open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CGM insulin bolus calculator arm (Experimental): All participants will receive the CGM insulin bolus calculator
  Interventions: Device: continuous glucose monitor based insulin bolus calculator

INTERVENTIONS:
Device: continuous glucose monitor based insulin bolus calculator — Participants will use the bolus calculator with meals to calculate their insulin bolus doses

SUMMARY:
This study examines the safety of an app-based insulin bolus calculator that utilizes glucose values from a continuous glucose monitor

DETAILED DESCRIPTION:
Individuals with type 1 diabetes and those with type 2 diabetes who are prescribed bolus insulin must decide on an insulin dose for any given meal. This dose is often based on what they are eating and their glucose value. Insulin bolus calculators may be helpful in recommending an insulin dose. This study examines the safety of an app-based insulin calculator manufactured by Welloc (Columbia, MD). This app uses the glucose value and trend arrow, in certain circumstances, to recommend a bolus insulin dose. This study is a single arm trial where continuous glucose monitoring metrics such as time in range will be measured before and after the study participants are given the app.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* type 2 diabetes
* using Dexcom G6 CGM system
* injecting bolus insulin

Exclusion Criteria:

* pregnancy,
* insulin pump use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
time in range | 30 days
  time in range using the calculator app will be non-inferior to baseline time in range

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Aleppo, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No